CLINICAL TRIAL: NCT06706141
Title: The Effect of Breast Cancer and Breast Self-Examination Health Education on Awareness, Beliefs and Practices Given to Female Students At the Faculty of Health Sciences of a University in Mogadishu, Somalia
Brief Title: The Effect of Breast Cancer and Breast Self-Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Eylul Yesilyurt, RN, Yüksek Lisans, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Recep Tayyip Erdoğan Faculty
Record Dates: First submitted 2024-11-17; First posted 2024-11-26 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Breast Carcinoma
Keywords: Awareness; Belief; Breast cancer; Breast self-examination; Health education; Students; Somalia
MeSH Terms: conditions — Breast Neoplasms; Breast Self-Examination; Health Education | interventions — Health Belief Model

STUDY DESIGN:
Intervention Model Description: A single-blind, randomized, controlled pretest-posttest experimental design was used for this research.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group received various interventions such as group education based on the health belief model, individual counseling, and brochures on screening. The training was given by two study team members in the faculty's conference hall, in the form of a presentation, discussion, and question-answer sessions, with the experimental group divided into two groups, lasting approximately 90 minutes. It was completed in 3 sessions with breaks every 30 minutes. For training hours, free hours when students did not have classes were chosen. For each training group, a member of the study team first gave a presentation on breast cancer and breast screening behaviors and BSE (30 minutes). Then, a film was shown on the BSE practice recommended by the World Health Organization (20 minutes) and training was given on how to perform correct and effective BSE on the breast model (20 minutes).
  Interventions: Behavioral: PowerPoint presentation.
- Control Group (No Intervention): The intervention group within the control group received health education on early diagnosis and prevention of breast cancer once the program was finished for them and all data had been gathered for both groups.

INTERVENTIONS:
Behavioral: PowerPoint presentation. — The training included topics such as breast anatomy; breast cancer incidence in Somalia, mortality, morbidity rates; breast cancer risk factors, importance of screening methods; The messages on breast self-examination, health belief models, breast cancer awareness, confidence for BSE, and perceived barriers/benefits for BSE were presented in a PowerPoint presentation. The procedure for performing breast self-examination was described using the English edition of Bristol-Myers Squibb Oncology. In the movie, BSE was made simpler with schematics showing the breast area that needed to be covered. Simple directions on which fingers to use and how to move them over the breast were provided. After the film, the emphasis shifted to helping students gain more self-assurance in their ability to accurately complete each BSE step. Students were encouraged to use proper palpation technique to find lumps by performing a breast examination on a silicone breast model.
  Other Names: The messages on breast self-examination, health belief models, breast cancer awareness, confidence for BSE, and perceived barriers/benefits for BSE were presented in a PowerPoint presentation.
  Arms: Experimental Group

SUMMARY:
Background: Somali women face extremely high mortality and incidence rates for breast cancer (BC). One of the suggested techniques for screening for breast cancer early detection is breast self-examination, or BSE. Studies have revealed that Somalian women, however, lack sufficient understanding and practice about BC and BSE. In this study, female students at a university in Mogadishu, Somalia, had their knowledge, attitudes, health beliefs, and BSE practices evaluated with reference to the effects of health belief model-based health education addressing BC and BSE.

Methods: It was conducted as a randomized controlled study on 86 female university students in Mogadishu, Somalia, between September 2021 and June 2022. Randomization was used to assign participants to the intervention group (n = 43) and control group (n = 43). Data were gathered using two instruments: a self-administered questionnaire was the first tool used to gather information on individuals' sociodemographic and level of awareness about BC and BSE. The health belief model scale is the second instrument. A validated checklist and a modified structured questionnaire were used to gather data. Subsequently, the students in the experimental group took part in the three 90-minute training sessions that made up the program. The control group did not receive any intervention. Three months later, further student data were gathered. Data analysis was performed using IBM-SPSS software version 20, descriptive and inferential statistical tests (T-test, chi-square, repeated measures).

ELIGIBILITY:
Inclusion Criteria:

* Turkish and Somali instructors work together at the faculty and students are given education in Turkish. If students are successful in one year of Turkish preparation, they can then continue to the department of their choice. The population of the research consisted of 500 female students over the age of 18 studying at the Recep Tayyip Erdoğan Faculty of Health Sciences in Mogadishu, Somalia.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female students
Enrollment: 86 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
post intervention | 3 months
  After the training, a post-test was administered to the experimental and control groups. Data were collected with "Sociodemographic Questionnaire", "Champion's health Belief Model Scale". Sociodemographic Questionnaire: This survey includes questions such as the age of the students, the education level of the mother and father, family income level, and family history of breast cancer. There were also 7 questions about students' breast cancer and breast self-examination. Champion's health Belief Model Scale: The 42-item Champion Health Belief Model Scale (CHBMS) was refined in subsequent research (1993, 1997, 1999) and was created by Victoria Champion in 1984 to assess women's attitudes and beliefs regarding breast cancer and breast self-examination. CHBMS has 6 subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want to share

REFERENCES:
- [Background] Altunkurek SZ, Hassan Mohamed S. Determine knowledge and belief of Somalian young women about breast cancer and breast self-examination with champion health belief model: a cross-sectional study. BMC Med Inform Decis Mak. 2022 Dec 8;22(1):326. doi: 10.1186/s12911-022-02065-4. PMID 36482433
- [Background] Yang S, Li P, Yu L, Liu N, Wang J, Guo P, Zhang X, Zhang W. Breast Cancer Awareness Based on Health Information Literacy and Influential Factors among Female Nursing Students in China. J Cancer Educ. 2022 Jun;37(3):546-554. doi: 10.1007/s13187-020-01844-9. PMID 32876864
- [Background] Andrew Tong JW, Hee MQ. The impact of an online educational game on breast cancer awareness among university female students, Malaysia: a pilot study. BMC Cancer. 2023 Oct 6;23(1):947. doi: 10.1186/s12885-023-11427-8. PMID 37803291
- See also: WHO — https://www.who.int/news-room/fact-sheets/detail/cancer
- See also: International Agency for Research on Cancer'na (IARC) — https://www.iarc.who.int/cancer-type/breast-cancer
- See also: Global Cancer Observatory (2022) — https://gco.iarc.who.int/media/globocan/factsheets/populations/706-somalia-fact-sheet.pdf.